CLINICAL TRIAL: NCT04299347
Title: Influence of the Restorative Cervical Margin Placement on the Supracrestal Tissue Attachment. A Longitudinal Study
Brief Title: Influence of the Restorative Cervical Margin Placement on the Supracrestal Tissue Attachment
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Professor, University of Siena
Other Study IDs: PR001
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Gingivitis
Keywords: subgingival restorations; proximal restorations; cytokine; biomarkers; GCF sampling
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid from the gingival sulcus
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the present study is to understand the influence that marginal/subgingival restorations exert on the surrounding periodontal tissues. Even though proximal restorations are routine in everyday clinical practice, few information is available as to whether or not they may have a detrimental effect on the supracrestal tissue attachment.

ELIGIBILITY:
Inclusion Criteria:

* an age range 18-70 years
* a good general health
* the ability to understand the phases of the trial and to stick to them for the whole length of the study
* the ability of will to release a written informed consent
* presence of a marginal cavity or a 2mm subgingival cavity
* presence of a cavity subgingival > 2mm

Exclusion Criteria:

* PPD>4mm
* patients affected by active periodontal disease
* patients smoking more than 10 cigarettes/pipes per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients coming to the Endodontic and Restorative department of Policlinico le Scotte- Siena, when eligible, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing | 12 months
  bleeding from the gingival sulcus when probing

SECONDARY OUTCOMES:
radiographic distance from the caries/margin of the restoration to the bone crest | 12 months
  LInear measurement between the most apical level of the restoration to the bone crest

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy